CLINICAL TRIAL: NCT02454504
Title: Quality of Awakening and Impact on Cognitive Function After Administration of Sugammadex in Robotic Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, Dr, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 307.CI
Record Dates: First submitted 2015-05-06; First posted 2015-05-27 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Anesthesiology Management
Keywords: Sugammadex; Delayed Emergence from Anesthesia; Curare; Robotic Surgical Procedures
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

ARMS (2):
- sugammadex (Active Comparator): this arm will receive sugammadex at the end of the surgery
  Interventions: Drug: sugammadex
- neostigmine (Active Comparator): this arm will receive neostigmine at the end of the surgery
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: sugammadex
  Arms: sugammadex
Drug: Neostigmine
  Arms: neostigmine

SUMMARY:
With the aim of enhancing the quality of surgery, the robotic cystectomy is often conducted using continuous intravenous infusion of curare, which ensures maximum neuromuscular relaxation until the end of the intervention. Sugammadex, administered for the reversal of deep neuromuscular blocked, enable rapid awakening. Moreover, Sugammadex seems to have a positive effect also on the recovery of cognitive function, psychomotor coordination and mental ability, effects undocumented in Literature.

The aim of the investigators study was to assess whether the reversal with sugammadex after intraoperative continuous infusion of rocuronium, can improve the quality of awakening.

ELIGIBILITY:
Inclusion Criteria:

* ASA score ≤ III
* Patients underwent robotic cystectomy

Exclusion Criteria:

* Cerebrovascular disease
* BMI ≥ 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
average score obtained on awakening according to specific test | 16 months
  cognitive function as assessed by the Mini Mental State Exam; quality of awakening as assessed by the Observer's Assessment of Alterness/sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena Cancer Institute, Rome, RM, Italy